CLINICAL TRIAL: NCT01354275
Title: IVF/ICSI Outcomes of OCP Plus GnRH Agonist Protocol Versus OCP Plus GnRH Antagonist Fixed Protocol in Women With PCOS
Brief Title: In Vitro Fertilization Outcomes of Two Treatment Protocols in Women With Polycystic Ovary Syndrome
Acronym: PCOS and ivf
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: . The trial would be continued if there was a difference of ≥3 % between trial arms. However, the difference between ongoing pregnancy rates was <1 %
Sponsor: Bulent Haydardedeoglu (Other)
Responsible Party: Sponsor-Investigator, Bulent Haydardedeoglu, IVF/ICSI Outcomes of OCP Plus GnRH Agonist Protocol Versus OCP Plus GnRH Antagonist Fixed Protocol in Women With PCOS: A Randomized Controlled Trial, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: BH532008; KA04/104 (Other: Baskent University KA04/104)
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: PCOS GnRH Antagonist and GnRH Agonist IVF/ICSI Cycles
Keywords: PCOS; IVF/ICSI; Clinical Pregnancy rates; GnRH Antagonist; GnRH Agonist
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRH Agonist (Active Comparator): oral contraceptive pill and GnRH Agonist IVF/ICSI cycle
  Interventions: Other: To compare the IVF/ICSI outcomes of GnRH Antagonist cycle versus GnRH agonist cycle
- GnRH Agonist Arm (Active Comparator): Oral contraceptive pill and day 21 GnRH agonist began, Day 3 of menstruation 150 IU FSH will be started. If 3 or more follicle reach >17 mm hCG will be administered.
  Interventions: Other: To compare the IVF/ICSI outcomes of GnRH Antagonist cycle versus GnRH agonist cycle; Other: GnRH Antagonist

INTERVENTIONS:
Other: To compare the IVF/ICSI outcomes of GnRH Antagonist cycle versus GnRH agonist cycle — 150 IU FSH dose and OCP plus GnRH Agonist (long luteal) IVF/ICSI cycle and 150 IU FSH dose and OCP plus GnRH Antagonist (Fixed protocol) IVF/ICSI Cycle
Other: GnRH Antagonist — GnRH Antagonist cycle; 150 IU FSH and sixth day Antagonist will be administered
  Arms: GnRH Agonist Arm

SUMMARY:
Outcomes of IVF/ICSI cycles of women with PCOS undergoing Gonadotropin Releasing Hormone (GnRH) agonist and GnRH Antagonist fixed protocol.

DETAILED DESCRIPTION:
Women with PCOS undergoing IVF/ICSI cycles will be evaluated by two different protocols. One arm of the study includes oral contraceptive plus GnRH agonist protocol with 150 IU FSH (standard dose) and second arm includes oral contraceptive plus GnRH Antagonist with 150 IU FSH dose and fixed 6th day starting of GnRH Antagonist.

ELIGIBILITY:
Inclusion Criteria:

* PCOS women undergoing ICSI cycles
* All women will be administered 150 IU rec FSH

Exclusion Criteria:

* Women having other endocrinopathies
* women older than 35
* third IVF/ICSI cycles
* previous and current use of metformin

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | March 2009 to June 2011
  Ongoing pregnancy rates measured in OCP plus GnRH Agonist and OCP plus GnRH Antagonist cycles in women with PCOS
clinical pregnancy rate | from march 2009 to july 2011
  To evaluate the clinical pregnancy rates of both study arms
Total gonadotropin use | From march 2009 to June 2011
  Total gonadotropin use of both study arms

SECONDARY OUTCOMES:
OHSS rates | from march 2009 to july 2011
  OHSS rates in both study groups
Total ongoing pregnancy rate | from march 2009 to june 2011
  Total ongoing pregnacy rates of per protocol group including freezing-thawing embryo transfer cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Haydardedeoglu, M.D., Study Chair — Baskent University
Locations (1):
- Bulent Haydardedeoglu, Adana, Turkey (Türkiye)